CLINICAL TRIAL: NCT05980637
Title: Effectiveness and Safety of Shaoyao Gancao Decoction With Addition on the Sleep-related Leg Cramps: A Randomized, Double-Blinded, Placebo-Controlled Trial
Brief Title: Effectiveness and Safety of Shaoyao Gancao Decoction With Addition on the Sleep-related Leg Cramps
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, Prof. Lin Zhixiu, Professor, Chinese University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Sleep-related Leg Cramps study
Record Dates: First submitted 2023-07-21; First posted 2023-08-08 (Actual); Last update posted 2023-08-08 (Actual); Status verified 2023-07

CONDITIONS: Sleep-related Leg Cramps
Keywords: Sleep-related Leg Cramps; Shaoyao Gancao Decoction with Addition
MeSH Terms: interventions — shaoyao gancao decoction

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Shaoyao Gancao Decoction with Addition (Active Comparator): 11g of Shaoyao Gancao Decoction with Addition granules twice daily for 4 weeks
  Interventions: Drug: Shaoyao Gancao Decoction with Addition
- Placebo (Placebo Comparator): 11g of placebo granules twice daily for 4 weeks
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Shaoyao Gancao Decoction with Addition — 11g twice daily for 4 weeks
  Other Names: SGDA
  Arms: Shaoyao Gancao Decoction with Addition
Other: Placebo — 11g twice daily for 4 weeks
  Arms: Placebo

SUMMARY:
A randomized, double-blinded, placebo-controlled clinical trial using a Chinese Medicine formula in treating Sleep-related Leg Cramps. Subjects will be randomized into a treatment group or placebo group for 4 weeks, and then post-treatment visit at week 6 and week 8.

DETAILED DESCRIPTION:
The sleep-related leg cramps (SRLC), also called nocturnal leg cramps (NLC), is a sleep-related limb movement disorder in which painful contractions of the calf or foot muscles occur during sleep, thereby interrupting the patient's rest. It can happen at any ages, but is particularly prevalent among the elderly.

In Chinese medicine, leg cramps, first mentioned in the book of "Huangdi Neijing" (The Yellow Emperor's Cannon of Internal Classic), is characterized by muscular spasm and contracture of a limb resulting in difficulty in relaxation and movement. SRLC is an impediment disease caused by the invasion of wind-cold damp pathogens in the muscles and sinews, together with the dual deficiency of qi and blood that fails to nourish the muscles and sinews, leading to painful contraction of muscles.

Currently, no treatments have been proven both safe and effective for SRLC. Passive stretching and deep tissue massage, which are patient-controlled maneuvers on relieving muscle tension, are usually recommended despite limited proof of effectiveness.

Shaoyao Gancao Decoction was first introduced in the book of "Shang Han Lun" (Treatise on Cold Attack) written by the venerated Physician Zhang Zhongjing in the Eastern Han dynasty. It consists of two herbs, i.e., Paeoniae Radix Alba and Glycyrrhizae Radix et Rhizoma Praeparata Cum Melle, and has the therapeutic functions of moderating painful spasms and alleviating pain. It is commonly used in Chinese medicine practice for treating abdominal pain, lack of strength in walking, spasms of the calf muscles, and restless leg syndrome. Modern pharmacological studies showed that Shaoyao Gancao Decoction possesses anti-inflammatory, analgesic and antispasmodic effects. It has been shown that the use of Shaoyao Gancao Decoction could inhibit mechanical and thermal hyperalgesia in rats with chronic compressive injury.

In 2009, a prospective observational pilot study was conducted to evaluate the effectiveness and safety of modified Shaoyao Gancao Decoction on 30 eligible subjects with SRLC in a cohort study and the result is positive.

Based on the positive results of the pilot study, it shows that SGDA is a promising herbal treatment method for SRLC, and propose a randomized, double-blinded and placebo-controlled trial to scientifically determine the effectiveness and safety of this formula for the treatment of Shaoyao Gancao Decoction with Addition (SGDA) of SRLC. Subjects will be randomized into a treatment group or placebo group for 4 weeks, and then post-treatment visits at week 6 and week 8.

ELIGIBILITY:
Inclusion Criteria:

* Aged 60 or above of both genders;
* Complain of muscular spasm and contracture of the lower limb with difficulty in relaxation and movement at night;
* Meet the diagnostic criteria of The International Classification of Sleep Disorders (3rd Edition) for SRLC [2];
* Meet the syndrome differentiation of the blood stasis or blood deficiency in Traditional Chinese Medicine.
* Regular SRLC occurs at least once per week on average within past month;
* Numeric Pain Rating Scale (NPRS) ≥ 5; and
* Willing to provide written informed consent.

Exclusion Criteria:

* Known mental disorder or neurologic disorder;
* Known serious organic disease including severe cardiovascular disease, post-stroke depression, cancer and dementia,;
* Currently on anticoagulants, antiplatelet medications, hypnotics, anxiolytics, positive inotropic drugs, corticosteroids and estrogenic and testosterone which may interfere with the study medications.
* Impaired hematological profile and liver / renal function exceeds the upper limit of the reference value by 2 times;
* Known allergic to Chinese medicines; and
* Any contraindications for taking Chinese medicines in the opinion of the investigators;
* Known history of lower limb surgery;
* Known pregnant or breast-feeding.

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2023-09-01 (Estimated); Primary Completion 2025-02-28 (Estimated); Study Completion 2025-08-31 (Estimated)

PRIMARY OUTCOMES:
The change in the Visual Analogue Scale (VAS) of painfulness | week 4
  The VAS is a unidimensional measure of pain intensity which will be self assessed by subjects daily, with the scale of 0 (no pain) to 10 (worst imaginable pain).

SECONDARY OUTCOMES:
The change in the Visual Analogue Scale (VAS) of painfulness | week 2
  The VAS is a unidimensional measure of pain intensity which will be self assessed by subjects daily, with the scale of 0 (no pain) to 10 (worst imaginable pain).
The change in the Visual Analogue Scale (VAS) of painfulness | week 6
  The VAS is a unidimensional measure of pain intensity which will be self assessed by subjects daily, with the scale of 0 (no pain) to 10 (worst imaginable pain).
The change in the Visual Analogue Scale (VAS) of painfulness | week 8
  The VAS is a unidimensional measure of pain intensity which will be self assessed by subjects daily, with the scale of 0 (no pain) to 10 (worst imaginable pain).
The change in frequency of SRLC | week 2
  Frequency of SRLC will be recorded by subjects daily.
The change in frequency of SRLC | week 4
  Frequency of SRLC will be recorded by subjects daily.
The change in frequency of SRLC | week 6
  Frequency of SRLC will be recorded by subjects daily.
The change in frequency of SRLC | week 8
  Frequency of SRLC will be recorded by subjects daily.
The change in total duration of SRLC per week | week 2
  Duration of SRLC will be recorded by subjects daily.
The change in total duration of SRLC per week | week 4
  Duration of SRLC will be recorded by subjects daily.
The change in total duration of SRLC per week | week 6
  Duration of SRLC will be recorded by subjects daily.
The change in total duration of SRLC per week | week 8
  Duration of SRLC will be recorded by subjects daily.
The change in the Short Form 36 Health Survey Questionnaire (SF-36) score | week 2
  The SF-36 is a 36-item scale, which measures eight domains of health status: physical functioning; physical role limitations; bodily pain; general health perceptions; energy/vitality; social functioning; emotional role limitations and mental health. It will be self assessed by subjects.
  The scores are transformed to range from 0 (where the respondent has the worst possible health) to 100 (where the respondent is in the best possible health).
The change in the Short Form 36 Health Survey Questionnaire (SF-36) score | week 4
  The SF-36 is a 36-item scale, which measures eight domains of health status: physical functioning; physical role limitations; bodily pain; general health perceptions; energy/vitality; social functioning; emotional role limitations and mental health. It will be self assessed by subjects.
  The scores are transformed to range from 0 (where the respondent has the worst possible health) to 100 (where the respondent is in the best possible health).
The change in the Short Form 36 Health Survey Questionnaire (SF-36) score | week 6
  The SF-36 is a 36-item scale, which measures eight domains of health status: physical functioning; physical role limitations; bodily pain; general health perceptions; energy/vitality; social functioning; emotional role limitations and mental health. It will be self assessed by subjects.
  The scores are transformed to range from 0 (where the respondent has the worst possible health) to 100 (where the respondent is in the best possible health).
The change in the Short Form 36 Health Survey Questionnaire (SF-36) score | week 8
  The SF-36 is a 36-item scale, which measures eight domains of health status: physical functioning; physical role limitations; bodily pain; general health perceptions; energy/vitality; social functioning; emotional role limitations and mental health. It will be self assessed by subjects.
  The scores are transformed to range from 0 (where the respondent has the worst possible health) to 100 (where the respondent is in the best possible health).
The change in the Pittsburg Sleep Quality Index (PSQI) | week 2
  PSQI measures the quality and pattern of sleep in older adult by measuring seven domains in 19 questions, which will be self-assessed by subjects.The scoring is 0-3 on a Likert scale.
The change in the Pittsburg Sleep Quality Index (PSQI) | week 4
  PSQI measures the quality and pattern of sleep in older adult by measuring seven domains in 19 questions, which will be self-assessed by subjects.The scoring is 0-3 on a Likert scale.
The change in the Pittsburg Sleep Quality Index (PSQI) | week 6
  PSQI measures the quality and pattern of sleep in older adult by measuring seven domains in 19 questions, which will be self-assessed by subjects.The scoring is 0-3 on a Likert scale.
The change in the Pittsburg Sleep Quality Index (PSQI) | week 8
  PSQI measures the quality and pattern of sleep in older adult by measuring seven domains in 19 questions, which will be self-assessed by subjects.The scoring is 0-3 on a Likert scale.
The score of Patient Global Impression of Change (PGIC) | week 2
  PGIC is a self-reported measure which reflects a patient's impression on the efficacy of treatment. It is a 7-point scale detecting patient's rating on the overall improvement of treatment. The patient can rate from 1 (very much improved) to 4 (no change) to 7 (very much worse).
The score of Patient Global Impression of Change (PGIC) | week 4
  PGIC is a self-reported measure which reflects a patient's impression on the efficacy of treatment. It is a 7-point scale detecting patient's rating on the overall improvement of treatment. The patient can rate from 1 (very much improved) to 4 (no change) to 7 (very much worse).
The score of Patient Global Impression of Change (PGIC) | week 6
  PGIC is a self-reported measure which reflects a patient's impression on the efficacy of treatment. It is a 7-point scale detecting patient's rating on the overall improvement of treatment. The patient can rate from 1 (very much improved) to 4 (no change) to 7 (very much worse).
The score of Patient Global Impression of Change (PGIC) | week 8
  PGIC is a self-reported measure which reflects a patient's impression on the efficacy of treatment. It is a 7-point scale detecting patient's rating on the overall improvement of treatment. The patient can rate from 1 (very much improved) to 4 (no change) to 7 (very much worse).

CONTACTS AND LOCATIONS:
Overall Officials: Zhixiu Lin, PhD, Principal Investigator — Hong Kong Institute of Integrative Medicine
Locations (1):
- Hong Kong Institute of Integrative Medicine, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: No